CLINICAL TRIAL: NCT00944580
Title: A Phase 1 Study to Determine the Immunologic Effects of a MAGE- A1, MAGE- A3, NY-ESO-1 Vaccine in Patients With High Risk Neuroblastoma, Osteogenic Sarcoma, and Rhabdomyosarcoma
Brief Title: A Vaccine Study for High Risk Cancers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: unexpectedly low screening results leading to poor accrual
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 30761; PSHCI 09-033
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Neuroblastoma; Rhabdomyosarcoma; Osteogenic Sarcoma
Keywords: MAGE-A1; MAGE-A3; NY-ESO-1; antigen; vaccine; dendritic cells; immunohistochemistry; immunology
MeSH Terms: conditions — Neuroblastoma; Rhabdomyosarcoma; Osteosarcoma | interventions — MAGEA1 protein, human; MAGEA3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine Intervention (Experimental): MAGE-A1, MAGE-A3, and NY-ESO-1 Vaccine: A regimen of three vaccines every two weeks. Each vaccine will contain 3,000,000-5,000,000 peptide pulsed dendritic cells. Imiquimod, a topical cream, will be applied to the vaccination site before and after each vaccination.
  Interventions: Biological: MAGE-A1, MAGE-A3, and NY-ESO-1 Vaccine

INTERVENTIONS:
Biological: MAGE-A1, MAGE-A3, and NY-ESO-1 Vaccine — A regimen of three vaccines every two weeks. Each vaccine will contain 3,000,000-5,000,000 peptide pulsed dendritic cells. Imiquimod, a topical cream, will be applied to the vaccination site before and after each vaccination.

SUMMARY:
The purpose of this study is to determine the safety and immunological effects of a vaccine for people diagnosed with high risk neuroblastoma, osteogenic sarcoma, and rhabdomyosarcoma. It is hypothesized that this vaccine could reduce the incidence of relapse.

DETAILED DESCRIPTION:
MAGE -A1, MAGE- A3, and NY-ESO-1 are antigens that can be found with significant frequency on neuroblastoma, rhabdomyosarcoma, and osteogenic sarcoma, three relatively common solid tumors that in some cases can be associated with a high risk for relapse. In this study each subject will be screened for the presence of these antigens, and an individualized vaccine will be developed and administered using the subject's own dendritic cells (DC).

This study consists of two phases: a screening phase and a treatment/vaccine phase. First, eligible individuals will be consented into the screening phase. Tumor specimens will be tested by immunohistochemistry or RT-PCR for the presence of MAGE- A1, MAGE- A3, and NY-ESO-1. Those testing positive for one or more antigen can be consented for the treatment phase of the study. Blood will be drawn for DC culture, and approximately one month later a series of three vaccines will be administered at two week intervals. Subjects will receive a topical medication called imiquimod to the vaccine site prior to and following each injection, to help immune cells travel into the area. Study participation occurs over 18 months and also involves periodic physical examinations and blood draws.

ELIGIBILITY:
Inclusion Criteria for Screening Phase:

Patient 1 to 70 years of age with neuroblastoma, rhabdomyosarcoma, or osteogenic sarcoma, who have one or more of the following high risk features:

* Neuroblastoma:

  * Stage IV disease
  * Stage III disease with n-myc amplification
* Osteogenic sarcoma:

  * Presence of metastases
  * Elevated alkaline phosphatase or LDH at diagnosis
  * Primary tumor affecting the axial skeleton
  * Poor histopathological response after completion of pre-surgical chemotherapy (≥10% viable tumor)
* Rhabdomyosarcoma:

  * Stage IV disease
  * Alveolar histology
  * Positive tumor margins, with lymph node positivity

Inclusion Criteria for Vaccine Phase:

* Patient meets all screening criteria and tumor is positive for NY-ESO-1, MAGE- A1, or MAGE-A3 by immunohistochemistry or RT-PCR.
* Patients who are between 3 months and 2 years following the completion of therapy, and have achieved at least a very good partial response to primary therapy.
* No chemotherapy is planned for one month following the last vaccination.
* Bilirubin <2 mg/dL, and SGOT/SGPT <2.5 x normal
* Creatinine clearance > 50ml/min as estimated by patient's serum creatinine, weight, and age
* Room air pulse oximetry >94%
* Patient is not pregnant
* Male and female sexually active patients of reproductive who wish to participate must agree to use acceptable contraception
* Patient is not moribund and has a projected life expectancy >6 months
* Lansky performance scale > 70, ECOG < 2 (Appendix I)
* Potential subjects will be tested for HIV 1 and 2 antibodies, HTLV 1/2 antibodies, and for HIV 1, hepatitis C and hepatitis B virus by NAT testing. - -Subjects testing positive for any of these pathogens will be ineligible for vaccine.
* White blood cells ≥ 2.5 K/µL, Hemoglobin ≥ 8 g/dL, Hematocrit > 25%, and Platelets ≥ 70 K/µL
* Patient does not have central nervous system involvement.
* Patient does not a have a history of autoimmune disease, specifically inflammatory bowel disease, systemic lupus erythematosis, or rheumatoid arthritis
* Patient is not receiving concurrent systemic steroid therapy
* Patient does not have a known systemic hypersensitivity to imiquimod or any vaccine component

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine if there is an amplification or new development of NY-ESO-1, MAGE-A1, or MAGE-A3 specific CD4+ or CD8+ T cells post-vaccination. | 2 years

SECONDARY OUTCOMES:
The investigators will determine the safety of vaccine and imiquimod administration in these patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G. Lucas, MD, Study Chair — Milton S. Hershey Medical Center